CLINICAL TRIAL: NCT05414539
Title: A Multicomponent Intervention to Rehabilitate Cognitive Impairment in People Post-stroke: Single-arm Feasibility Study
Brief Title: OptiCogs: A Multicomponent Intervention to Rehabilitate Cognitive Impairment in People Post-stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Limerick (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: OptiCogs
Record Dates: First submitted 2022-02-21; First posted 2022-06-10 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-02

CONDITIONS: Stroke, Cardiovascular; Cognitive Impairment
Keywords: Feasibility; Stroke; Cognitive impairment; Multicomponent rehabilitation
MeSH Terms: conditions — Myocardial Infarction; Cognitive Dysfunction; Stroke

STUDY DESIGN:
Intervention Model Description: A non-randomised single-arm feasibility study using a pre-test: post-test design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): OptiCogs Online is a 6-week telehealth intervention consisting of cognitive, physical activity and educational components. Cognitive component of the intervention: Throughout the six-week intervention period, there will be three individualised one-to-one cognitive sessions (occurring on week one, week three and week five), delivered by an occupational therapist. Physical activity: The physical activity component will be delivered via telehealth by a physiotherapist.
  * Aerobic: Progressions from Week 1-Week 6 will result in individual achieving 60 mins moderate intensity aerobic activity @ frequency of 3 times per week as tolerated.
  * Muscular strengthening: Progressions from Week 1-Week 6 will result in the person post-stroke achieving 10 strengthening exercises x 10 reps x 3 sets @ frequency of 3 times per week as tolerated. Cognitive education: The cognitive education component is underpinned by the Bridges stroke self-management package and based on self-efficacy principles.
  Interventions: Other: OptiCogs Online

INTERVENTIONS:
Other: OptiCogs Online — A multicomponent intervention to rehabilitate cognitive deficits in people post-stroke

SUMMARY:
OptiCogs Online is a complex multicomponent intervention comprising of cognitive, physical activity and educational components.

DETAILED DESCRIPTION:
OptiCogs Online was developed in accordance with the MRC framework for the development and evaluation of complex interventions. Given the known interactions and interconnectivity of cognitive domains required for optimal cognitive functioning post-stroke, a systematic review of 64 studies addressing all types of non-pharmacological rehabilitation interventions which may improve multiple cognitive domains in people post-stroke was conducted. Within this review, rehabilitation interventions were categorised as multicomponent interventions, physical activity interventions, cognitive rehabilitation interventions, NIBS protocols, occupational-based interventions and other interventions. The most consistent evidence in our systematic review and meta-analysis supported multicomponent interventions, with significant improvement demonstrated for general cognitive function and memory outcomes. Specifically, multicomponent interventions wherein a form of cognitive rehabilitation was conducted in conjunction with a form of physical activity were shown to improve cognitive functioning in people post-stroke.

As well as meta-analytic evidence, we drew from qualitative findings which explored the perspectives of PpS, caregivers and healthcare professionals on the design and delivery of an intervention to improve cognitive functioning in PpS. Qualitative findings and input from clinical experts emphasised the importance of information provision, peer support and meaningful engagement. As such, each component of OptiCogs Online is supplemented with an educational or 'cognitive education' session wherein group discussion covers different aspects of cognitive functioning. As well as drawing on findings from our qualitative study, this 'cognitive education' component is underpinned by the Bridges stroke self-management package and based on self-efficacy principles.

To this end, a complex multicomponent intervention comprising of cognitive, physical activity and educational components was developed in line with the MRC framework.

ELIGIBILITY:
Inclusion Criteria:

* People with a physician-confirmed diagnosis of stroke. Stroke may be ischaemic or haemorrhagic in nature.
* People aged ≥18 years old; with confirmed mild to moderate cognitive impairment using the Oxford Cognitive Screen (OCS) (in accordance with cut-offs for impairment for OCS-plus subtasks (Demeyere et al. 2021a) and the Addenbroke's Examination III (ACE III) with a cut-off score of 88/100 (Takenoshita et al. 2019).
* People post-stroke who have a Modified Rankin Scale (MRS) score of 0-3
* Capacity to provide informed consent
* People post-stroke who are able to express their basic needs, verbally or not
* Have access to a smartphone, laptop or tablet with an internet connection
* Willingness/ interest in participating in an online intervention
* Physician-confirmed suitability to partake in this intervention

Exclusion Criteria:

* Physician-confirmed contraindications for undertaking physical activity e.g., safety, presence of unstable heart disease
* People with diagnosed TIA will be excluded
* People post-stroke with known active delirium or dementia will be excluded
* People post-stroke with a diagnosis of known pre-stroke cognitive impairment
* People post-stroke with moderate or severe visuospatial neglect

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-05-09 (Actual); Primary Completion 2022-06-24 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | 6 weeks
  The proportion of participants who are recruited to the study.
Adherence rate | 6 weeks
  The proportion of participants who adhere to the treatment protocol of 6 weeks. We will determine the level of adherence to the intervention protocol using the self-report diary.
Adverse events | 6 weeks
  Number of participants with adverse events as a measure of safety. Adverse events include a fall, illness, medical complication etc.
Acceptability of OptiCogs Online | 6 weeks
  The proportion of participants reporting that OptiCogs Online is acceptable. Acceptability (satisfaction) of the OptiCogs intervention will be assessed using a self-report questionnaire developed by the researchers containing 5-point Likert scales: 1= "strongly disagree"; 2= "disagree"; 3= "neutral"; 4= "agree"; 5= "strongly agree".
Retention rate | 6 weeks
  The proportion of participants who are lost to follow-up

SECONDARY OUTCOMES:
Oxford Cognitive Screen-plus (OCS-plus) | 6 weeks
  Changes in cognitive function from pre-intervention to post-intervention in accordance with the cut-offs for impairment for OCS-Plus subtasks.
Addenbrooke's Cognitive Assessment (III) ACE (III) | 6 weeks
  Changes in cognitive function from pre-intervention to post-intervention in accordance with ACE III score out of 100.
Fatigue severity scale (FSS) | 6 weeks
  ). The FSS is a 9-item scale which measures the severity of fatigue and its effect on ADLs on a 7-point scale. The FSS is shown as a valid and reliable measure of fatigue in people post-stroke
PROMIS-10 Physical Functioning | 6 weeks
  • Physical function (PF) will be assessed using a physical functioning subset of the patient reported outcomes measurement information system (PROMIS) scale.
Stroke Specific Quality of Life Scale | 6 weeks
  • Mood and social participation will be assessed using the relevant subscales of the Stroke-Specific Quality of Life Scale-12 (SSQoL-12).

CONTACTS AND LOCATIONS:
Overall Officials: Sara Hayes, PhD, Principal Investigator — University of Limerick
Locations (1):
- University of Limerick, Limerick, Ireland

REFERENCES:
- [Derived] O' Donoghue M, Boland P, Taylor S, Hennessy E, Murphy E, Leahy S, McManus J, Lisiecka D, Purtill H, Galvin R, Hayes S. OptiCogs: feasibility of a multicomponent intervention to rehabilitate people with cognitive impairment post-stroke. Pilot Feasibility Stud. 2023 Oct 18;9(1):178. doi: 10.1186/s40814-023-01300-7. PMID 37853485